CLINICAL TRIAL: NCT04840056
Title: Prediction of Gastric Cancer in Intestinal Metaplasia and Atrophic Gastritis - Application of Artificial Intelligence in Histology and Clinical Data
Brief Title: Prediction of Gastric Cancer in Intestinal Metaplasia and Atrophic Gastritis
Acronym: GIMA
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: 2021.082
Record Dates: First submitted 2021-03-23; First posted 2021-04-09 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Intestinal Metaplasia; Atrophic Gastritis
Keywords: artificial intelligence
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intestinal Metaplasia: patient with history of histologically proven gastric intestinal metaplasia
- Atrophic gastritis: patient with history of histologically proven atrophic gastritis

SUMMARY:
The primary objectives of this study are:

* To identify clinical or histological factors associated with gastric cancer development in patients with IM and AG
* To establish a machine learning algorithm for prediction of future gastric cancer risks and individual risk stratification in patient with IM and AG

DETAILED DESCRIPTION:
This is a two-part retrospective study including a clinical data part and a pathology part. A training cohort will be developed from approximately 70% of included cases. It will be followed by a validation cohort with the remaining cases.

Clinical data will be collected retrospectively using the Clinical Data Analysis and Reporting System (CDARS) and Clinical management System (CMS). A cluster-wide cohort (New Territories East Cluster, NTEC) consisting of patients with history of histologically-proven gastric IM and AG will be identified and included for subsequent analysis. The data collection period for the retrospective data will be 2000-2020.

Histology slides will be retrieved retrospectively when available (within NTEC). Whole slide imaging technique will be utilized for the development of training and validation cohorts with machine learning algorithms in the pathology part.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years of age
* Histologically proven atrophic gastritis or intestinal metaplasia (at antrum and/or body and/or angular of stomach)

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinical data will be collected retrospectively using the Clinical Data Analysis and Reporting System (CDARS) and Clinical management System (CMS). A cluster-wide cohort (New Territories East Cluster, NTEC) consisting of patients with history of histologically-proven gastric IM and AG will be identified and included for subsequent analysis. The data collection period for the retrospective data will be 2000-2020.
  Histology slides will be retrieved retrospectively when available (within NTEC). Whole slide imaging technique will be utilized for the development of training and validation cohorts with machine learning algorithms in the pathology part.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer and gastric dysplasia | 20 years
  The primary endpoint is the incidence of gastric cancer (intestinal-type) and gastric dysplasia (low grade and high grade dysplasia).

SECONDARY OUTCOMES:
Overall accuracy of machine learning model | 20 years
  Overall accuracy of machine learning models will be evaluated
Sensitivity of machine learning model | 20 years
  Sensitivity of machine learning model will be evaluated
Specificity of machine learning model | 20 years
  Specificity of machine learning model will be evaluated
Positive predictive value of machine learning model | 20 years
  Positive predictive value of machine learning model will be evaluated
Negative predictive value of machine learning model | 20 years
  Negative predictive value of machine learning model will be evaluated
Area under the receiver operating characteristic curve of machine learning model | 20 years
  Area under the receiver operating characteristic curve of machine learning model will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers